CLINICAL TRIAL: NCT02992340
Title: A Multicentre, Phase 1B/2 Study of Varlitinib in Combination With Gemcitabine and Cisplatin for Treatment naïve Advanced or Metastatic Biliary Tract Cancer.
Brief Title: Varlitinib in Combination With Gemcitabine and Cisplatin for Treatment naïve Advanced or Metastatic BTC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to terminate the study and not proceed to Phase 2.
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-007
Record Dates: First submitted 2016-12-08; First posted 2016-12-14 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2020-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1B (Experimental): Varlitinib (starting dose at 200 mg BID) Cisplatin Gemcitabine
  Interventions: Drug: Varlitinib; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Varlitinib — Per oral (PO) Varlitinib BID (starting dose at 200 mg BID)
  Other Names: ASLAN001
Drug: Cisplatin — On D1 and D8, every 3 weeks. Cisplatin (25 mg per square meter of body surface area) in 1 litre of 0.9% saline with 20 mmol of potassium chloride and 8 mmol of magnesium sulfate intravenous (IV) infusion for 2 hours, followed by 500 mL of 0.9% saline over 30 minutes before the administration of Gemcitabine
Drug: Gemcitabine — On D1 and D8, every 3 weeks. Gemcitabine (1000 mg per square meter of body surface area) as a 30-minute infusion.

SUMMARY:
The study intends to evaluate the following objectives in patients with advanced or metastatic biliary tract cancer who have not received systemic therapy for advanced/metastatic disease.

Primary Objectives:

Phase 1B

* To determine the maximum tolerated dose (MTD), as determined by dose-limiting toxicities (DLTs), and to characterise the safety profile of Varlitinib in combination with Gemcitabine and Cisplatin.

Phase 2A

* To further evaluate the safety and tolerability of Varlitinib in combination with Gemcitabine and Cisplatin at the recommended phase 2 dose (RP2D).
* To provide a preliminary assessment of the clinical activity of Varlitinib in combination with Gemcitabine and Cisplatin at the RP2D as measured by Objective Response Rate (ORR) and progression-free survival (PFS) (based on RECIST v1.1)

Phase 2B

* To compare the efficacy of Varlitinib in combination with Gemcitabine and Cisplatin to placebo in combination with Gemcitabine and Cisplatin as measured by progression-free survival (based on RECIST v1.1).

DETAILED DESCRIPTION:
In phase 1B part, patients will receive Varlitinib plus Gemcitabine and Cisplatin, and follow a modified 3+3+3 study dose escalation scheme starting from Varlitinib 200 mg BID. The primary objective of the phase 1B part is to determine the MTD of Varlitinib when given in combination with Gemcitabine and Cisplatin, and to characterise the safety profile of the study treatment regimen.

Based on the determined MTD and clinical information obtained from phase 1B part of the study, the DSMB will review the safety data and other clinical data, together with the sponsor, determine the MTD as well as the recommended phase 2 dose (RP2D). The sponsor will make a decision when to proceed with the phase 2A part of the study.

The phase 2A part of the study is designed as a single arm expansion, enrolling a further 20 patients at the RP2D. The purpose of the phase 2A expansion study is to confirm the safety and tolerability of the RP2D in a larger number of patients, and to provide preliminary estimates of the clinical activity of Varlitinib in combination with Gemcitabine and Cisplatin, prior to embarking on the larger, randomised phase 2B part of the trial.

The phase 2B part will be a two-arm, double-blinded, placebo controlled study. Patients will be randomised into 2 arms to receive Varlitinib plus Gemcitabine and Cisplatin, or placebo plus Gemcitabine and Cisplatin. The primary endpoint of the phase 2B part is progression-free survival (PFS). The randomisation will be stratified by primary tumour location (gall bladder or non-gall bladder).

Patient screening activities including informed consent and study eligibility verification will be performed within 21 days prior to first dose of the study medication. Radiological imaging to assess the disease status will be performed at baseline and every 6 weeks from Cycle 1 Day 1. Blood samples will be taken during the screening phase, treatment period until end of treatment. Patients will be required to complete safety follow-up within 28 days after the last administration of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of respective country's legal age or older at the time of written informed consent.
2. Patient must be able to understand and willing to provide informed consent for participation in the study and donation of tumour tissue (archival or fresh) for evaluation of relevant exploratory endpoints.
3. Patient must have histologically or cytologically confirmed advanced (unresectable) or metastatic biliary tract cancer, including intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer, or carcinoma of the Ampulla of Vater, with no prior systemic therapy for advanced/metastatic disease. This includes clinical diagnosis of biliary tract cancer with histological confirmation of adenocarcinoma.
4. For phase 1B and 2A only: Presence of radiologically measured disease with at least one, not previously irradiated, measurable lesion according to RECIST v.1.1.
5. No evidence of clinically significant biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below or equal to 1.5 x upper level of normal (ULN).
6. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Patient with adequate organ and haematological function prior to first dose of study medication:

   a. Haematological function, as follows: i. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L ii. Platelet count ≥ 100 x 109/L iii. Haemoglobin level ≥ 10 g/dl b. Renal functions, as follows: i. Serum creatinine ≤ 1.5x ULN or eGFR > 60 ml/min/1.73m2 c. Hepatic function, as follows: i. Total bilirubin ≤ 1.5 x ULN ii. AST and ALT ≤ 5 x ULN

Exclusion Criteria:

1. Patients with radiation or local treatment 6 weeks prior to screening for the target lesion(s).
2. Patients with major surgical procedures within 21 days prior to screening.
3. Patients with known brain metastases.
4. Patients with malabsorption syndrome, diseases significantly affecting gastrointestinal function, resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications which in the opinion of the Investigator could jeopardize the validity of the study results. Any extent of stomach resection will be excluded.
5. Pre-existing peripheral sensory neuropathy ≥ grade 2 according to CTCAE (v.4.03).
6. Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, diabetes, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients with any history of other malignancy unless in remission for more than 1 year prior to screening (Non-melanoma skin carcinoma and carcinoma-in-situ of uterine cervix treated with curative intent is not exclusionary).
8. Patients with a known history of HIV, decompensated cirrhosis, HCV infection, and for phase 1B: HBV infection with detectable HBV deoxyribonucleic acid (DNA) or abnormal transaminase; for phase 2A & 2B: HBV infection with HBV DNA exceeding 2000 IU/mL.
9. Any history or presence of clinically significant cardiovascular, respiratory, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease or any other condition, which, in the opinion of the investigator, could jeopardise the safety of the patient or the validity of the study results.
10. Patients with known history of drug addiction within last 1 year.
11. Patients who may need continuous treatment with proton pump inhibitors or strong CYP3A4 inhibitors during the study period.
12. Female patients who are pregnant or breast-feeding.
13. Patients who have received any investigational drug (or have used an investigational device) within the last 14 days before receiving the first dose of study medication.
14. Patients who have received immunotherapy for cancer, including but not limited to immune checkpoint inhibitors, monoclonal antibody, cancer vaccine, and cell therapy.
15. Patient with unresolved or unstable serious toxicity (≥ CTCAE 4.03 Grade 2) from prior administration of another investigational drug and/or prior cancer treatment.
16. Have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis, or have a history of interstitial lung disease or current interstitial lung disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Phase 1B: Maximum tolerated dose (MTD) of Varlitinib | DLT period is 3 weeks
  To determine the maximum tolerated dose (MTD), as determined by dose-limiting toxicities (DLTs), and to characterise the safety and tolerability profile of Varlitinib as determined by the adverse events in combination with Gemcitabine and Cisplatin.
Phase 1B: Safety and toxicity | Through study duration, estimated 3 years
  Determined by the adverse events.
Phase 2A: Safety and tolerability | Through study duration, estimated 3 years
  Determined by adverse events
Phase 2A: Safety and tolerability | Through study duration, estimated 3 years
  Determined by safety parameters (including vital signs, ECG parameters, clinical laboratory tests)
Phase 2A: Safety and tolerability | Through study duration, estimated 3 years
  Other measures of tolerability such as dose interruptions, treatment exposure and dose intensity.
Phase 2A: Objective Response Rate (ORR) | Through study duration, estimated 3 years
  ORR is defined as the number (%) of patients with at least one visit response of CR or PR. Data obtained up until the earlier of progression or the last evaluable assessment prior to starting subsequent therapy, will be included in the assessment of ORR.
Phase 2A: Progression Free Survival (PFS) | Through study duration, estimated 3 years
  PFS is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression). Progression is defined in accordance with the RECIST v1.1 criteria and will be derived programmatically.
Phase 2B: Progression Free Survival (PFS) | Through study duration, estimated 3 years
  PFS is defined as the time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression). Progression is defined in accordance with the RECIST v1.1 criteria and will be derived programmatically based on data from the Independent Central Review (ICR) of radiological data.

SECONDARY OUTCOMES:
Objective Response Rate (ORR)(Phase 1B) | Through study duration, estimated 3 years
  ORR is defined as the number (%) of patients with at least one visit response of CR or PR. Data obtained up until the earlier of progression or the last evaluable assessment prior to starting subsequent therapy, will be included in the assessment of ORR.
Objective Response Rate (Phase 2B) | Through study duration, estimated 3 years
  ORR is defined as the number (%) of patients with at least one visit response of CR or PR. Data obtained up until progression or the last evaluable assessment in the absence of progression, will be included in the assessment of ORR.
Disease control rate (DCR) (Phase 1B, Phase 2A and Phase 2B) | Through study duration, estimated 3 years
  DCR is defined as the number (%) of patients with at least one visit response of CR or PR, or with stable disease for a minimum of twelve weeks (- 5 days) from randomisation (Phase 2B) or starting treatment (Phase 1B and Phase 2A). For Phase 2B, data obtained up until progression, or last evaluable assessment in the absence of progression, will be included in the assessment of DCR.
Duration of response (DoR) (Phase 1B, Phase 2A and Phase 2B) | Through study duration, estimated 3 years
  DoR is defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression.
Overall Survival (OS) (Phase 2A and Phase 2B only) | Through study duration, estimated 3 years
  OS is defined as time from the start of treatment (Phase 2A) or randomisation (Phase 2B) until death by any cause.
Incidence of AEs (Phase 2B) | Through study duration, estimated 3 years
  Changes from baseline in safety parameters (including vital signs, ECG parameters, clinical laboratory tests) as categorized in accordance to CTCAE v4.03
Pharmacokinetics of Varlitinib (Phase 1B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Maximum plasma concentration (Cmax)
Pharmacokinetics of Varlitinib (Phase 1B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Time to Cmax (tmax)
Pharmacokinetics of Varlitinib (Phase 1B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Area under the plasma concentration-time curve from 0 to 6 hours (AUC0-6), and area under the plasma concentration-time curve from 0 to 12 hours (AUC0-12).
Pharmacokinetics of Varlitinib (Phase 1B) | Cycle 2 Day 1
  Pre-dose concentration (Ctrough)
Pharmacokinetics of Varlitinib (Phase 1B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Accumulation ratio of AUC0-6 (Day 22) compared to AUC0-6 (Day 1) (RacAUC0-6), accumulation ratio of AUC0-12 (Day 22) compared to AUC0-12 (Day 1) (RacAUC0-12)
Pharmacokinetics of Varlitinib (Phase 1B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Accumulation ratio of Cmax (Day 22) compared to Cmax (Day 1) (RacCmax).
Pharmacokinetics of Varlitinib (Phase 1B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Accumulation ratio of Cmax (Day 22) compared to Cmax (Day 1) (RacCmax)
Pharmacokinetics of Varlitinib (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Maximum plasma concentration (Cmax)
Pharmacokinetics of Varlitinib (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Time to Cmax (tmax)
Pharmacokinetics of Varlitinib (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Area under the plasma concentration-time curve from 0 to 6 hours (AUC0-6), and area under the plasma concentration-time curve from 0 to 12 hours (AUC0-12)
Pharmacokinetics of Varlitinib (Phase 2B) | Cycle 2 Day 1
  Pre-dose concentration (Ctrough)
Pharmacokinetics of Varlitinib (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Accumulation ratio of AUC0-6 (Day 22) compared to AUC0-6 (Day 1) (RacAUC0-6), accumulation ratio of AUC0-12 (Day 22) compared to AUC0-12 (Day 1) (RacAUC0-12)
Pharmacokinetics of Varlitinib (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Accumulation ratio of Cmax (Day 22) compared to Cmax (Day 1) (RacCmax)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Maximum plasma concentration (Cmax)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Time to Cmax (tmax)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Last measurable concentration (Clast)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Terminal half-life (t1/2)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Mean residence time (MRT)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Volume of distribution at the terminal phase (Vz) and volume of distribution at the steady-state (Vss)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Plasma clearance (Cl)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Area under the plasma concentration-time curve from 0 to t (AUC0-t), and area under the plasma concentration-time curve from 0 to infinite (AUC0-inf)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Accumulation ratio of AUC0-inf (Day 22) compared to AUC0-inf (Day 1) (RacAUC0-inf)
Pharmacokinetics of Gemcitabine, dFdU (gemcitabine metabolite) and Cisplatin (Phase 2B) | Cycle 1 Day 1 and Cycle 2 Day 1
  Accumulation ratio of Cmax (Day 22) compared to Cmax (Day 1) (RacCmax)

CONTACTS AND LOCATIONS:
Overall Officials: ASLAN Pharmaceuticals ASLAN Pharmaceuticals, Study Director — contact@aslanpharma.com
Locations (3):
- Singapore, Singapore
- Seoul, South Korea
- Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No